CLINICAL TRIAL: NCT02769351
Title: A Multicentre, Prospective Registry to Evaluate the Safety and Efficacy of Minimally Invasive Ultrafiltration Treatment and Its Effect on Symptoms and Rehospitalisation in Patients With Advanced Volume Overload
Brief Title: Global rEgistry on decongestioN Therapy Using Less invasivE UltraFiltration
Acronym: GENTLE-UF
Status: Terminated | Type: Observational
Why Stopped: It was decided to prematurely terminate the GENTLE-UF registry as a parallel study conducted with the same device has been prematurely terminated due to low recruitment.
Sponsor: Fresenius Medical Care Deutschland GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: UF-HF-01-INT; DRKS00009836 (Registry Identifier: DRKS: German Clinical Trials Register)
Record Dates: First submitted 2016-03-21; First posted 2016-05-11 (Estimated); Results first posted 2021-07-08 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-04

CONDITIONS: Acute Heart Failure; Cardiac Decompensation; Volume Overload
Keywords: volume overload; heart failure; cardiac decompensation; ultrafiltration
MeSH Terms: conditions — Heart Failure; Edema | interventions — Ultrafiltration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- periph. minimal invasive ultrafiltration: Patients with volume overload receiving ultrafiltration
  Interventions: Device: periph. minimal invasive ultrafiltration

INTERVENTIONS:
Device: periph. minimal invasive ultrafiltration — ultrafiltration via a peripheral single-needle
  Other Names: ultrafiltration

SUMMARY:
In patients with advanced volume overload, minimally invasive ultrafiltration treatment in the acute phase can have a positive effect on clinical outcome. The aim is to collect treatment data in the context of a prospective registry of the safety and performance of minimally invasive ultrafiltration. The data will be recorded via an electronic case report form (eCRF); the eCRF runs on a server located in Germany and complies with current data protection regulations. It is intended to include about 300-500 patients with advanced volume overload at a minimum of 10 sites. In addition, data on a disease management programme (in-body measurement and home monitoring) will be recorded in up to 40 of these patients. The treatment data from each patient will be recorded over 12 months. An interim analysis will be performed after 150 patients have been observed for 6 months. The knowledge about ultrafiltration in volume overload obtained from the registry, in some cases in combination with a disease management programme, is intended to improve the body of evidence. In addition, the data will be used for hypothesis generation.

DETAILED DESCRIPTION:
There may be various reasons why an increased accumulation of fluid occurs in tissue. The most common causes include heart failure, kidney failure or cirrhosis of the liver. In rare cases, oedema can develop following septicaemia. The usual treatment of oedema involves diuretics, i.e. water tablets, which remove excess fluid from the body and which can be administered either orally or intravenously. For some years now, it has also been possible to use ultrafiltration to treat oedema. This involves filtering and removing excess fluid from the blood. This individual method enables a precisely defined amount of fluid to be withdrawn. Access to the blood circulation is usually via a central venous catheter, as in acute dialysis. Current international treatment guidelines recommend that consideration should be given to ultrafiltration therapy in the context of treatment of diuretic-resistant volume overload (e.g. second- or third-line therapy for acute decompensated heart failure). There are, however, to date no clinical data on a combined treatment regimen of diuretics and supportive ultrafiltration. Accordingly, ultrafiltration may be included in clinical guidelines either only with a low level of evidence (e.g. IIb in the ACCF/AHA guidelines) or not at all (ESC guidelines). The main reasons for the limited body of evidence for ultrafiltration are, on the one hand, the invasive nature of the usual procedures (these usually require the insertion of a central venous catheter) and structural barriers in the health system (ultrafiltration is normally offered by nephrologists and not by cardiologists). With an increasing clinical need and limited medical alternatives, particularly in view of the frequently occurring diuretic resistance in heart failure, there is an urgent medical need to fill this gap in evaluation evidence. In the context of the registry, the CHIARA system, a minimally invasive (i.e. via a peripheral venous access) extracorporeal ultrafiltration system, is used for the treatment of decompensated volume overload. The CHIARA system has a CE mark for the intended purpose of ultrafiltration of the blood of patients suffering from heart failure, acute or chronic renal failure or excess body fluid. It is planned to use the medical device in connection with this intended purpose only. In participating hospitals, patients will be treated with this new treatment strategy of minimally invasive ultrafiltration treatment in support of diuretic drug therapy in the acute phase of volume overload. It is possible with the use of ultrafiltration therapy to control volume overload and reduce it on an individual basis, so that diuretics can be given sparingly and, as a consequence, diuretic resistance and a deterioration of renal function due to diuretic uptitration can be avoided.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years
* Inpatient-treated patients with acute volume overload, preferably in association with cardiac decompensation with signs of incipient diuretic resistance (lack of increase in urine output despite significant escalation of diuretic therapy; e.g. ≥80 mg furosemide / 24 h or less than 1375 mL urine output/40 mg furosemide per 24 h or equivalent dose of other loop diuretics [established clinically or from the medical history])
* New York Association Functional Class (NYHA) III-IV at inclusion
* Systolic or diastolic cardiac dysfunction (HF-REF or HF-PEF)
* Adequate venous access (preferably peripheral arm vein) allowing a flow rate ≥ 60 mL / min
* Written consent to the use of data in the registry (where necessary, by a legal guardian).

Exclusion Criteria:

* Contraindication to anticoagulation (e.g. known heparin-induced thrombocytopenia, severe bleeding)
* Terminal renal failure (stage V, GFR <15 mL)
* Cardiogenic shock, e.g. in association with acute coronary syndrome (ACS)
* Other diseases or factors that, in the study doctor's opinion, constitute a potential contraindication to ultrafiltration
* Pregnant women, women in labour, breast-feeding women or women of childbearing potential, who are without adequate contraception or are planning a family. NB: a pregnancy test is performed systematically in women of childbearing age and the patient is not included in the event of pregnancy (positive test). It is absolutely essential that women, who have a negative test and who are included in the study, have an effective contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with minimally invasive ultrafiltration in support of diuretic drug therapy in the acute phase of volume overload.
Sampling Method: Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2015-12-03 (Actual); Primary Completion 2019-03-04 (Actual); Study Completion 2019-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henning T Baberg, MD, Principal Investigator — Helios Klinikum Berlin Buch, Berlin
Locations (19):
- Germany (11):
  - Universitätsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Helios Klinik für Herzchirurgie GmbH Karlsruhe, Karlsruhe, Baden-Wurttemberg
  - Universitätsklinikum Mannheim, Mannheim, Baden-Wurttemberg
  - Klinikum Stuttgart, Stuttgart, Baden-Wurttemberg
  - Städtisches Klinikum Braunschweig, Braunschweig, Lower Saxony
  - Helios Klinikum Hildesheim, Hildesheim, Lower Saxony
  - Uniklinik RWTH Aachen, Aachen, North Rhine-Westphalia
  - Helios Klinik Attendorn, Attendorn, North Rhine-Westphalia
  - Helios Klinikum Duisburg, Duisburg, North Rhine-Westphalia
  - HELIOS Klinikum Erfurt, Erfurt, Thuringia
  - Helios Klinikum Berlin Buch, Berlin
- Sweden (6):
  - Falun Hospital, Falun
  - SUS Skanes University Hosptal, Malmo
  - University Hospital Örebro, Örebro
  - Karolinska University Hospital, Stockholm
  - Danderyd University Hospital, Stockholm
  - Uppsala University Hospital, Uppsala
- Switzerland (2):
  - Kantonsspital Aarau, Aarau
  - UniversitätsSpital Zurich, Zurich

IPD SHARING:
Plan to Share IPD: No
Overall results will be published. Individual participant data will not be made available.

REFERENCES:
- [Background] Yancy CW, Jessup M, Bozkurt B, Butler J, Casey DE Jr, Drazner MH, Fonarow GC, Geraci SA, Horwich T, Januzzi JL, Johnson MR, Kasper EK, Levy WC, Masoudi FA, McBride PE, McMurray JJ, Mitchell JE, Peterson PN, Riegel B, Sam F, Stevenson LW, Tang WH, Tsai EJ, Wilkoff BL; American College of Cardiology Foundation; American Heart Association Task Force on Practice Guidelines. 2013 ACCF/AHA guideline for the management of heart failure: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2013 Oct 15;62(16):e147-239. doi: 10.1016/j.jacc.2013.05.019. Epub 2013 Jun 5. No abstract available. PMID 23747642
- [Background] McMurray JJ, Adamopoulos S, Anker SD, Auricchio A, Bohm M, Dickstein K, Falk V, Filippatos G, Fonseca C, Gomez-Sanchez MA, Jaarsma T, Kober L, Lip GY, Maggioni AP, Parkhomenko A, Pieske BM, Popescu BA, Ronnevik PK, Rutten FH, Schwitter J, Seferovic P, Stepinska J, Trindade PT, Voors AA, Zannad F, Zeiher A; Task Force for the Diagnosis and Treatment of Acute and Chronic Heart Failure 2012 of the European Society of Cardiology; Bax JJ, Baumgartner H, Ceconi C, Dean V, Deaton C, Fagard R, Funck-Brentano C, Hasdai D, Hoes A, Kirchhof P, Knuuti J, Kolh P, McDonagh T, Moulin C, Popescu BA, Reiner Z, Sechtem U, Sirnes PA, Tendera M, Torbicki A, Vahanian A, Windecker S, McDonagh T, Sechtem U, Bonet LA, Avraamides P, Ben Lamin HA, Brignole M, Coca A, Cowburn P, Dargie H, Elliott P, Flachskampf FA, Guida GF, Hardman S, Iung B, Merkely B, Mueller C, Nanas JN, Nielsen OW, Orn S, Parissis JT, Ponikowski P; ESC Committee for Practice Guidelines. ESC guidelines for the diagnosis and treatment of acute and chronic heart failure 2012: The Task Force for the Diagnosis and Treatment of Acute and Chronic Heart Failure 2012 of the European Society of Cardiology. Developed in collaboration with the Heart Failure Association (HFA) of the ESC. Eur J Heart Fail. 2012 Aug;14(8):803-69. doi: 10.1093/eurjhf/hfs105. No abstract available. PMID 22828712

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Out of 104 patients recruited, 46 patients have been included in the safety population (SP; all patients included in analysis), and 44 patients have been included in the analysis population (AP; patients included in analysis with at least one ultrafiltration treatment).
Period: Overall Study
Arm/Group | Periph. Minimal Invasive Ultrafiltration
Started | 46 (SP)
Completed | 4 (SP)
Not Completed | 42

BASELINE CHARACTERISTICS:
Population: Baseline characteristics have been analyzed based on the analysis population.
Arm/Group | Periph. Minimal Invasive Ultrafiltration
Number analyzed (Participants) | 44
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Baseline characteristics have been analyzed based on the analysis population.However, due to the observational character of the study, data are not always available for all patients. The actual number of patients with available data is depicted per variable.
  years
    number analyzed (Participants) | 42
    (all) | 74.71 (10.76)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Baseline characteristics have been analyzed based on the analysis population.However, due to the observational character of the study, data are not always available for all patients. The actual number of patients with available data is depicted per variable.
  Participants
    number analyzed (Participants) | 42
    Female | 14
    Male | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Weight, Continuous [Mean (Standard Deviation); unit: kg] — Population: Baseline characteristics have been analyzed based on the analysis population.However, due to the observational character of the study, data are not always available for all patients. The actual number of patients with available data is depicted per variable.
  kg
    number analyzed (Participants) | 42
    (all) | 90.19 (21.16)
Height, Continuous [Mean (Standard Deviation); unit: cm] — Population: Baseline characteristics have been analyzed based on the analysis population.However, due to the observational character of the study, data are not always available for all patients. The actual number of patients with available data is depicted per variable.
  cm
    number analyzed (Participants) | 41
    (all) | 171.93 (10.30)
Body-Mass-Index (BMI), Continuous [Mean (Standard Deviation); unit: kg/m^2] — Population: Baseline characteristics have been analyzed based on the analysis population.However, due to the observational character of the study, data are not always available for all patients. The actual number of patients with available data is depicted per variable.
  kg/m^2
    number analyzed (Participants) | 41
    (all) | 30.03 (5.10)

OUTCOME MEASURES:

1. Primary Outcome: Rehospitalisation (Yes/no) Due to Exacerbation of Heart Failure/Volume Overload of Other Origin
Description: The number of rehospitalizations due to heart failure resp. volume overload has been measured as a clinical endpoint and analyzed based on the AP.
Time Frame: 12 months
Population: The outcome has been analyzed based on the AP (44 patients).
Measure: Number; unit: Rehospitalizations
Arm/Group | Periph. Minimal Invasive Ultrafiltration
Number analyzed (Participants) | 44
Rehospitalizations
  Rehospitalization due to Heart Failure | 7
  Rehospitalization due to other reasons | 12

2. Secondary Outcome: Significant Deterioration of Kidney Function - Creatinine
Description: Significant deterioration of kidney function has been measured as a safety endpoint and analyzed based on the SP. The variables have been measured at recruitment, discharge from the index hospitalization, Outpatient visit I (3-9 months) and Outpatient visit II (12 months).
Time Frame: Recruitment; Discharge from Index Hospitalization; Outpatient visit I (3-9 months); Outpatient visit II ( 12 months)
Population: The outcome has been analyzed on the SP (46 patients). However, due to the observational character of the study, data are not always available for all patients. The actual number of patients with available data is depicted per time point.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Periph. Minimal Invasive Ultrafiltration
Number analyzed (Participants) | 46
mg/L
  Creatinine at Recruitment: number analyzed (Participants) | 40
  Creatinine at Recruitment | 208.30 (71.79)
  Creatinine at Discharge from Index Hospitalization: number analyzed (Participants) | 32
  Creatinine at Discharge from Index Hospitalization | 180.66 (78.13)
  Creatinine at Outpatient visit I: number analyzed (Participants) | 9
  Creatinine at Outpatient visit I | 224.99 (162.7)
  Creatinine at Outpatient visit II: number analyzed (Participants) | 3
  Creatinine at Outpatient visit II | 430.31 (454.01)

3. Secondary Outcome: Significant Deterioration of Kidney Function - Urea
Description: as for outcome 2
Time Frame: Recruitment; Discharge from Index Hospitalization; Outpatient visit I (3-6 months); Outpatient visit II (12 months)
Population: The outcome has been analyzed on the SP (46 patients). However, due to the observational character of the study, data are not always available for all patients. The actual number of patients with available data is depicted per time point and variable.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Periph. Minimal Invasive Ultrafiltration
Number analyzed (Participants) | 46
mg/dL
  Urea at Recruitment: number analyzed (Participants) | 28
  Urea at Recruitment | 21.7 (15.01)
  Urea at Discharge from Index Hospitalization: number analyzed (Participants) | 25
  Urea at Discharge from Index Hospitalization | 51.67 (168.40)
  Urea at Outpatient visit I: number analyzed (Participants) | 3
  Urea at Outpatient visit I | 282.99 (457.51)
  Urea at Outpatient visit II: number analyzed (Participants) | 0

4. Secondary Outcome: Significant Deterioration of Kidney Function - eGFR (Estimated Glomerular Filtration Rate)
Description: as for outcome 2
Time Frame: Recruitment, Discharge from index hospitalization, Outapteint visit I (3-6 months), Outpatient visit II (12 months)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mL/min*1.73^2
Arm/Group | Periph. Minimal Invasive Ultrafiltration
Number analyzed (Participants) | 46
mL/min*1.73^2
  eGFR at Recruitment: number analyzed (Participants) | 40
  eGFR at Recruitment | 28.58 (15.56)
  eGFR at Discharge from Index hositalization: number analyzed (Participants) | 33
  eGFR at Discharge from Index hositalization | 37.82 (24.48)
  eGFR at Outaptient visit I: number analyzed (Participants) | 9
  eGFR at Outaptient visit I | 36.19 (30.87)
  eGFR at Outpatient visit II: number analyzed (Participants) | 3
  eGFR at Outpatient visit II | 41.52 (52.96)

5. Secondary Outcome: Significant Deterioration of Kidney Function - Cystatin
Description: as for outcome 2
Time Frame: recruitment, discharge from the index hospitalization, Outpatient visit I (3-9 months), Outpatient visit II (12 months)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/mL
Arm/Group | Periph. Minimal Invasive Ultrafiltration
Number analyzed (Participants) | 46
mg/mL
  Cystatin at Recruitment: number analyzed (Participants) | 5
  Cystatin at Recruitment | 2.26 (1.72)
  Cystatin at Discharge from index Hospitalization: number analyzed (Participants) | 2
  Cystatin at Discharge from index Hospitalization | 0.09 (0.13)
  Cystatin at Outpatient visit I: number analyzed (Participants) | 0
  Cystatin at Outpatient visit II: number analyzed (Participants) | 1
  Cystatin at Outpatient visit II | 6.99

ADVERSE EVENTS:
Time Frame: Adverse events were collected from signing the informed consent up to 12 month after recruitment.
Description: Adverse Event Definition has been done according to a form based on ISO 14155
Arm/Group | Periph. Minimal Invasive Ultrafiltration
All-Cause Mortality (participants affected / at risk) | 15/46
Serious Adverse Events (participants affected / at risk) | 22/46
Other Adverse Events (participants affected / at risk) | 4/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Periph. Minimal Invasive Ultrafiltration (N=46)
Cardiac failure (Cardiac disorders) | 9 (10)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 2 (2)
Fluid retention (Metabolism and nutrition disorders) | 1 (1)
Hospitalisation (Surgical and medical procedures) | 2 (2)
Death (General disorders) | 4 (4)
Staphylococcal sepsis (Infections and infestations) | 2 (2)
Cardiomyopathy (Cardiac disorders) | 1 (1)
Palliative care (Surgical and medical procedures) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Catheter placement (Surgical and medical procedures) | 1 (1)
Peritoneal catheter insertion (Surgical and medical procedures) | 1 (1)
Demyelinating polyneuropathy (Immune system disorders) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Periph. Minimal Invasive Ultrafiltration (N=46)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Thrombosis in device (Product Issues) | 1 (1)
Hospitalisation (Surgical and medical procedures) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-22): https://cdn.clinicaltrials.gov/large-docs/51/NCT02769351/Prot_SAP_000.pdf